CLINICAL TRIAL: NCT04582422
Title: Exploring Preschool Children the Use of Interventional Touch Therapy in the Treatment of Children's Dental Clinics Reducing Medical Fearing Randomized Controlled Trials
Brief Title: Interventional Touch Therapy in the Treatment of Children's Dental Clinics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NYMUH-IRB No. 2020B001
Record Dates: First submitted 2020-05-07; First posted 2020-10-09 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-10

CONDITIONS: Dental Fear; Nursing
Keywords: Touch therapy; Fear

STUDY DESIGN:
Intervention Model Description: Interventional research
Who Masked: Outcomes Assessor
Masking Description: Single blinding
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Touch Therapy (Experimental): The main purpose is to provide "Touch Therapy" intervention measures, the degree of fear of dental treatment for preschool children.
  Use the chip chip tool (PCT) to ask the children's degree of fear of dental treatment. The control group uses questionnaires to ask the caregiver's age, social and economic status, education, past dental experience, etc. In the intervention group, the questionnaire was used to ask the caregiver's age, socioeconomic status, education, past dental experience, etc. During the waiting process, first follow the touch flow chart and perform the touch in the waiting area for 10 minutes. When visiting the treatment chair, the companion will be asked to touch the child's unilateral hand for 5 minutes during the consultation process. A small chair is provided to accompany the child for a total of 15 minutes. The two groups will use the chip tool again after the consultation , Ask the children how scared they are after seeing a doctor,
  Interventions: Other: Touch Therapy"
- dental education (No Intervention): The Chip Chip Tool (PCT) asked the children how scared they were about dental visits. The control group used questionnaires to ask the caregiver 's age, socioeconomic status, education, past dental experience, etc. before the visit to provide routine dental care, provide dental health education, how to use toothbrush Dental floss education,

INTERVENTIONS:
Other: Touch Therapy" — During the waiting process, first follow the touch flow chart and perform the touch in the waiting area for 10 minutes. When visiting the treatment chair, the companion will be asked to touch the child's unilateral hand for 5 minutes during the consultation process. A small chair is provided to accompany the child for a total of 15 minutes. The two groups will use the chip tool again after the consultation
  Arms: Touch Therapy

SUMMARY:
This study mainly wants to discuss the anxiety and fear of children's dental visits. For preschool children, separation anxiety can be obvious at this time. The main research is 1. To explore the degree of fear of dental visits in preschool children;2. Children who are touched therapy, there differences in fear of children 's dental treatment? If parents or important others can provide touching care to increase children 's sense of safety, reduce children 's fear of dental visits, and improve the quality of dental care The main purpose of the study.

DETAILED DESCRIPTION:
In this study, a parallel randomized study design was adopted. The intervention of the experimental group was a "Touch Therapy " measure. The control group To provide dental health education in accordance with the routine procedures of children's dental visits, how to use toothbrushes, dental floss education, a total of 90 samples were collected. Children who meet the inclusion criteria of this study are randomly assigned to the experimental group and the control group. The main purpose is to provide "Touch Therapy " intervention measures, and the difference in fear of dental treatment for preschool children.

Use the chip chip tool (PCT) to ask the children's degree of fear of dental treatment. The control group uses questionnaires to ask the caregiver's age, social and economic status, education, past dental experience, etc. In the intervention group, the questionnaire was used to ask the caregiver's age, socioeconomic status, education, past dental experience, etc. During the waiting process, first follow the touch flow chart and perform the touch in the waiting area for 10 minutes. When visiting the treatment chair, the companion will be asked to touch the child's unilateral hand for 5 minutes during the consultation process. A small chair is provided to accompany the child for a total of 15 minutes. The two groups will use the chip tool again after the consultation , Ask the children how scared they are after seeing a doctor, submit the collected data to a third party for analysis, and design a single-blind study.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged three to six who are admitted to the dental clinic.
2. Children and their families can communicate in Taiwanese and have a clear awareness and a digital concept.

Exclusion Criteria:

1. Children with cognitive developmental delay or visual impairment and hearing impairment.
2. Children who need to use a protective restraint board if they cannot cooperate with the medical treatment at this time.
3. The children in the control group actively need others to provide touch for more than 2 minutes due to their needs.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2021-06-25 (Actual); Study Completion 2021-06-25 (Actual)

PRIMARY OUTCOMES:
Chinese chip tools worry about score differences | Evaluation 20 minutes before a single dental treatment, 5 minutes after the intervention, and 5 minutes after the completion of the dental treatment
  Using the Chinese bargaining tool to compare the scores of "touch therapy" children and children receiving dental health education and guidance, different intervention measures affect the fear of dental treatment

SECONDARY OUTCOMES:
Demographic Research Questionnaire | Before dental treatment
  Parents' basic information includes gender, age, education, income, occupation, dental treatment experience, and children's basic information including gender, age, dental treatment experience, whether the child regularly uses fluoride, whether the child has dental caries in the past, using dental floss, using gargle Saliva, this dental treatment project

CONTACTS AND LOCATIONS:
Locations (1):
- NationalYMUH, Yilan, No.169, Siaoshe Rd, Taiwan

IPD SHARING:
Plan to Share IPD: No